CLINICAL TRIAL: NCT02506894
Title: Fetal Middle Cerebral Artery Doppler in Preterm Births Receiving Magnesium Sulfate for Neuroprotection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Abdel Fattah, assistant professor of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Mgso4 for neuroprotection
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- magnesium sulfate (Active Comparator): this group will receive magnesium sulfate loading dose 6 g in 500 cc of ringer solution over 20 minutes then maintenance dose of 1 g/ hour for 24 hours.
  Interventions: Drug: Magnesium Sulfate
- placebo group (Placebo Comparator): this group will receive sodium chloride 0.9% solution for 24 hours.
  Interventions: Other: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: Magnesium Sulfate — magnesium sulfate will be given for 24 hours
  Other Names: MgSO4
  Arms: magnesium sulfate
Other: 0.9% sodium chloride solution — normal saline will be given as intravenous drip over 24 hours
  Arms: placebo group

SUMMARY:
Two groups of women with preterm labor will be included. One will receive magnesium sulfate for neuroprotection and the other will receive placebo. Fetal middle cerebral artery Doppler indices will be measured before and after intake of either magnesium sulfate or placebo to find if any significant changes occur in fetal cerebral blood flow.

DETAILED DESCRIPTION:
The study will include women with preterm labor with gestational age less than 32 weeks. women will be randomized to receive either magnesium sulfate (loading dose 6 g over 20 minutes followed by maintenance dose of 1 g/hour for 24 hours), or placebo in the form of sodium chloride solution 0.9% over 24 hours. Fetal middle cerebral artery Doppler indices [Peak systolic velocity (PSV), Pulsatility index (PI), and resistance index (RI)] will be recorded before and after treatment in both groups. Results of Doppler indices will be compared between both groups and before and after intake of magnesium sulfate to find out if middle cerebral artery Doppler of the fetus can explain the mechanism behind the use of magnesium sulfate for fetal neuroprotection in preterm births.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with preterm labor
* gestational age less than 32 weeks
* singleton pregnancy

Exclusion Criteria:

* contraindication or hypersensitivity to magnesium
* preeclampsia
* multiple pregnancy
* intake of magnesium sulfate in this pregnancy before

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
changes in fetal middle cerebral artery Doppler indices | 3 months

SECONDARY OUTCOMES:
maternal adverse effects of magnesium sulfate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdel Fattah Abdel Moety, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt